CLINICAL TRIAL: NCT03531073
Title: A Multicentre Observational Psoriatic Arthritis Cohort Study Addressing Real-life Outcomes of a Treat to Target Approach in Routine Clinical Practice.
Brief Title: Multicentre ObservatioNal Initiative in Treat to Target Outcomes in Psoriatic Arthritis
Acronym: MONITOR
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 230600
Record Dates: First submitted 2018-02-08; First posted 2018-05-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Psoriatic Arthritis
Keywords: treat to target
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An optional substudy will collect biological samples for research purposes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Standard care cohort: This study is observational. Patients will receive standard treatment as given in usual clinical practice with no intervention as part of the study. As per current clinical practice guidelines and UK reimbursement rules for biologics in PsA, patients will receive a pragmatic treat to target approach using step up standard therapies. Patients will usually receive methotrexate first line, initially 15mg ow increasing to 25mg ow as tolerated. In case of non-response, an additional DMARD will be used (sulfasalazine up to 3g daily or leflunomide 20mg od). If two DMARDs are failed and patients are eligible for biologic therapy under UK National Institute of Health and Clinical Excellence (NICE) guidance, then biologics will be used.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — This study is observational and patients will receive treatment for their psoriatic arthritis as clinically indicated. As per standard practice in this observational cohort, patients are most likely to be treated with methotrexate as the most common first line therapy in PsA. This cohort is the basis of a TWiCs (Trials Within Cohorts) study design and interventional studies will be nested within this in future. Whilst the cohort will receive treatment for their PsA as part of their routine clinical care, this treatment will be decided according to routine care and not protocolised.

SUMMARY:
MONITOR is a cohort study recruiting patients with a new diagnosis of psoriatic arthritis (PsA) which will establish outcomes using a pragmatic feasible 'treat to target' approach in a real-life clinic population. It is the central cohort for a planned Trials Within Cohorts (TWiCs) design which will test alternative therapies and interventions in embedded clinical trials comparing outcomes to those receiving "standard care" in the cohort.

DETAILED DESCRIPTION:
Psoriatic Arthritis (PsA) is an inflammatory arthritis estimated to occur in 15% of people with psoriasis, affecting around 150,000 people in the United Kingdom (UK). The 2015 European League Against Rheumatism (EULAR) Treatment recommendations for PsA incorporating as its first recommendation that "treatment should be aimed at reaching the target of remission or, alternatively, minimal/low disease activity, by regular monitoring and appropriate adjustment of therapy". Despite the evidence and the EULAR recommendations supporting 'treat to target' in PsA, it has not been widely implemented due to concerns about feasibility and cost-effectiveness. This cohort will establish a pragmatic feasible 'treat to target' approach in a real-life clinic population which we believe can provide similar clinical and health-related quality of life outcomes.

The primary outcome will be the proportion of patients achieving a good response measured by the PsA Disease Activity Score (PASDAS) at 48 weeks. Additional domains including participation, fatigue and emotional wellbeing will be assessed for the first time. Finally the costs of this pragmatic intervention will be established using health economic analysis.All patients will receive treatment as usual following the current British Society of Rheumatology (BSR) and EULAR guidance as standard of care.

As a cohort for a "Trials within Cohorts" or TWiCs design, the patients consenting to participate will also be asked if they consent to be approached for future interventional trials linked to the cohort and whether they consent for their data to be used as a comparator in these future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female
* Aged 18 years or above.
* Clinical diagnosis of PsA based upon the Classification of PsA (CASPAR) criteria(23))
* Active PsA defined by ≥1 tender or ≥1 swollen joint or ≥1 enthesis (site of attachment of tendon to bone)
* Not previously received treatment with synthetic or biologic disease-modifying anti-rheumatic drugs (DMARDs) for their articular disease.
* In the Investigator's opinion, is able and willing to comply with all study requirements.

Exclusion Criteria:

* Current or previous treatment of arthritis with synthetic DMARDs (including methotrexate, leflunomide or sulfasalazine) or biologic DMARDs (including tumour necrosis factor (TNF), interleukin (IL)12/23 or IL17 inhibitor therapies) or targeted synthetic DMARDs (phosphodiesterase (PDE) 4 or Janus kinase (JAK) inhibitor therapies).
* Use of investigational therapies within 1 month or 5 biological half-lives of the baseline study visit(whichever is longer)
* Women who are pregnant, nursing or planning pregnancy during the following 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with psoriatic arthritis who have not previously had treatment with disease modifying therapy.
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Psoriatic arthritis disease activity score (PASDAS) | 48 weeks
  A composite measure of PsA disease activity. This score is a composite measure of disease activity in PsA. There is only one total score which ranges from 0-10 with higher numbers indicating more active disease. Low disease activity is defined as <3.2.

SECONDARY OUTCOMES:
Psoriatic Arthritis Impact of Disease (PsAID) | 48 weeks
  A questionnaire assessing the overall impact of disease on a patient. This is a scale of 12 questions (scored 0-10) which are combined with published weighting scales to one final 0-10 score where 0 is "no impact" and 10 is "maximal impact". There are no subscales. Patient acceptable symptom state is <=4.
Treatment satisfaction questionnaire for medications (TSQM) | 48 weeks
  A questionnaire assessing benefit and tolerability of the treatment given. There are 4 subscales measuring effectiveness (questions 1-3), side effects (questions 4-8), convenience (questions 9-11), and global satisfaction (questions 12-14). Each is scored 0-100 where 100 is good and 0 is bad. The subscales are not combined to one final score.
Healthcare costs | 48 weeks
  Healthcare costs of treatment given will be calculated for the patients within the cohort will be collected at 24 weeks and 48 weeks using self-reported questionnaires. The data collected will record indirect costs as well as direct non-medical costs. This is one measure that will report the healthcare costs for the patients in the cohort. This could be split into subscales of drug costs, healthcare provision costs and costs of investigations.
  Unit cost data will be obtained from national databases such as the British National Formulary (BNF) and Personal Social Services Research Unit (PSSRU) Costs of Health and Social Care.
Health related quality of life | 48 weeks
  HRQoL will be calculated using the EuroQol 5 dimension 5 level (EQ-5D-5L) questionnaire which is a generic measure of health related quality of life. This will be collected at baseline, 6 and 12 months and responses to the EQ-5D will be converted into multi-attribute utility scores using an established algorithm. Possible values range from -0.224 to 1 with 0 representing death, 1 representing full health and negative values representing states worse than death. Thus a higher score represents better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rombach I, Tillett W, Jadon D, Tucker L, Watson M, Francis A, Sinomati Y, Eldridge L, Dritsaki M, Dutton SJ, Al-Mossawi H, Gullick N, Thompson B, Coates LC. Treating to target in psoriatic arthritis: assessing real-world outcomes and optimising therapeutic strategy for adults with psoriatic arthritis-study protocol for the MONITOR-PsA study, a trials within cohorts study design. Trials. 2021 Mar 4;22(1):185. doi: 10.1186/s13063-021-05142-7. PMID 33663566